CLINICAL TRIAL: NCT04675931
Title: An Adaptive, Randomized, Active-controlled, Open-label, Sequential Cohort, Multicenter Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Intravenous Cipargamin (KAE609) in Adult and Pediatric Participants With Severe Plasmodium Falciparum Malaria (KARISMA - KAE609's Role In Severe Malaria)
Brief Title: To Evaluate Efficacy, Safety, Tolerability and PK of Intravenous Cipargamin in Participants With Severe Plasmodium Falciparum Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Wellcome Trust (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CKAE609B12201; 217692/Z/19/Z (Other Grant/Funding Number: Wellcome Trust and EDCTP within the PAMAFRICA Grant); 2020-005035-70 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Severe Malaria
Keywords: KAE609; cipargamin; artesunate; intravenous; i.v.; pediatric; dose-finding; safety; tolerability; pharmacokinetics
MeSH Terms: conditions — Malaria | interventions — NITD 609; Artesunate; Artemether, Lumefantrine Drug Combination; Artemether; Lumefantrine

STUDY DESIGN:
Intervention Model Description: This will be an adaptive, multicenter, randomized, open label, sequential cohort study in participants aged ≥ 12 years old in Cohorts 1-2 and < 12 years old to ≥ 6 months in Cohorts 3-5 with a diagnosis of moderately severe and severe P. falciparum malaria. In Cohorts 1-2, participants will get randomized to one of the three treatment arms (2 dose of intravenous cipargamin or intravenous artesunate - comparator ). After Cohort 2, interim analysis will be performed to take one best dose of intravenous cipargamin forward for Cohorts 3-5. Participants in Cohorts 3-5 with be randomized to one of two treatments arms ( intravenous cipargamin or intravenous artesunate - comparator).
Who Masked: Outcomes Assessor
Masking Description: Although the study is open label however in order to minimize the potential impact of treatment knowledge, treatment allocation, dose information, PK/AAG assessment schedule and concentration data, as well as other data that may result in systematic unblinding will not be available to the Clinical Trial Team (CTT) (particularly clinicians, trial statisticians, trial programmers) until the database is locked after IA of Cohorts 1-2. After interim database lock, the CTT would be unblinded with the results, however, the blinding will then be continued for Cohorts 3-5 until the final database is locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- IV KAE609 Dose regimen 1 (Experimental): Intravenous KAE609 (cipargamin) 20 mg
  Interventions: Drug: KAE609
- IV KAE609 Dose regimen 2 (Experimental): Intravenous KAE609 (cipargamin) 40 mg
  Interventions: Drug: KAE609
- IV KAE609 Dose regimen 3 (Experimental): Intravenous KAE609 (cipargamin) Dose regimen 3 (dose will be evaluated post Interim analysis from Cohort 1 and Cohort 2.
  Interventions: Drug: KAE609
- IV Artesunate (Active Comparator): IV Artesunate 2.4 mg/kg (for participants weighing at least 20 kg) IV Artesunate 3 mg/kg (for participants weighing less than 20 kg)
  Interventions: Drug: IV Artesunate
- Coartem (Other): Standard of care (Coartem) will be given to all participants for 3 days as part of treatment.
  Interventions: Drug: Coartem

INTERVENTIONS:
Drug: KAE609 — Two doses of Intravenous Cipargamin will be evaluated in the initial phase of the study (Cohorts 1-2).
  These doses will cover a wider exposure range and facilitate the selection of an appropriate dose for later Cohorts 3-5.
  Other Names: Cipargamin
  Arms: IV KAE609 Dose regimen 1; IV KAE609 Dose regimen 2; IV KAE609 Dose regimen 3
Drug: IV Artesunate — Parenteral artesunate is the WHO recommended first line treatment for severe malaria. Hence IV artesunate is used as comparator. Also, this will be used as rescue medication for participants where IV KAE609 is not working.
  Other Names: Artesunate
  Arms: IV Artesunate
Drug: Coartem — Oral Standard of Care
  Other Names: Artemether; Lumefantrine
  Arms: Coartem

SUMMARY:
The purpose of this study is to identify the safe and effective dose of intravenous cipargamin in participants with moderately severe and severe malaria.

The study also intends to evaluate clinical treatment success using a novel clinical endpoint for drug development in severe malaria.

Severe malaria is a medical emergency and is affecting primarily young children in Africa. Injectable artesunate is the standard of care for the treatment of severe malaria and is highly efficacious. However, the spread of artemisinin-resistance in Plasmodium falciparum in Asian countries poses a threat for future treatment of patients with this life-threatening disease. To mitigate this risk, there is a need of another drug in malaria endemic countries. Cipargamin treatment results in rapid clearance of parasites including artemisinin resistant parasites.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Participants aged ≥ 12 years with moderately severe malaria as defined in (prostration and/or repeated vomiting) without presence of other signs of severe malaria (and with high P. falciparum parasitemia (60,000-250,000 parasites per µl)

  * Subsequent Cohorts 2 to 5: Participants diagnosed with severe malaria as defined in modified version of WHO criteria and P. falciparum parasite count of ≥ 5000 per µl
  * Cohort 2: Participants aged ≥ 12 years
  * Cohort 3: Participants aged 6 - < 12 years
  * Cohort 4: Participants aged 2 - < 6 years
  * Cohort 5: Participants aged ≥ 6 months - < 2 years

Exclusion Criteria:

Exclusion criteria applying to all Cohorts 1 to 5:

* Mixed Plasmodium infections
* Treatment with quinine or artemisinin derivative or any other antimalarial drug or any antibiotic with known antimalarial activity within 12 hours of screening.
* Signs/symptoms of severe malnutrition in general accordance with WHO guidelines:

  1. Under 18 years: <-3 Z-scores of WHO growth standard for weight-for-height/length (in children < 5 years) or BMI for age (5-18 years), or very low mid-upper arm circumference (MUAC < 115 mm in children < 12 years, < 160mm 12-18 years), or bilateral pitting edema
  2. Over 18 years: BMI < 16 kg/m2 or MUAC < 160mm or bilateral pitting edema
* Known underlying illness, surgical or medical condition, which is not related to ongoing event of severe malaria and which might jeopardize the participant's health in case of participation in the study or which might alter the distribution, metabolism or excretion of study treatment. For example:

  1. neurological or neurodegenerative disorders,
  2. cardiac, renal, or hepatic disease, diabetes,
  3. epilepsy, cerebral palsy,
  4. known or suspected to be HIV-1 positive and/or receiving antiretroviral treatment
  5. malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
  6. known or suspected cases of active infections or concurrent febrile illness such as TB, Typhoid, COVID-19 etc.

Additional exclusion criteria are as follows:

Exclusion criteria for Cohort 1:

* ALT > 5 x the upper limit of normal range (ULN), regardless the level of total bilirubin
* Total bilirubin is > 3 mg/dL
* Body weight of < 35 kg or >75 kg

Exclusion criteria for Cohort 2:

* Body weight of < 35 kg or >75 kg
* Participants diagnosed as moderately severe malaria due to repeated vomiting without presence of any of the symptoms of severe malaria

Exclusion criteria for Cohorts 3 to 5:

* Body weight of < 5 kg
* Participants diagnosed as moderately severe malaria due to repeated vomiting without presence of any of the symptoms of severe malaria

Ages: 6 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Percentage of participants achieving at least 90% reduction in Plasmodium falciparum (P. falciparum) at 12 hours | Day 1 (12 Hours)
  A blood draw will be performed at each collection time point for parasitemia assessment.

SECONDARY OUTCOMES:
Percentage of participants achieving clinical success over time | Day 3 (48 Hours), Day 4 to Day 29
  Clinical success is a composite endpoint based on following criterias:
  1. Is participant dead or alive
  2. Presence of asexual parasites (yes/no)
  3. Presence of any of the key signs of severe malaria (yes/no)
Percentage of participants with individual signs of severe malaria over time | Day 1 to Day 29
  Individual signs of severe malaria over time will be monitored for the presence of the following signs of severe malaria during the entire study duration:
  1. Altered consciousness - Prostration or GCS < 11 for participants > 5 years / BCS < 3 for participants =< 5 years of age
  2. Renal Impairment - Serum creatinine > 3xULN or > 3 mg/dL or need for renal replacement therapy
  3. Acidosis - Serum lactate > 4 mmol/L
  4. Respiratory distress - present or absent
  5. Severe anemia - Hb < 5 g/dl or Hb < 7g/dl in pediatric and adults respectively or need of blood transfusion
  6. Jaundice - Serum bilirubin > 3 g/dl
  7. Hypoglycemia- plasma glucose < 40 mg/dL
Percentage of participants developing hemolysis (early and delayed) after treatment | Day 8 and Day 29
  Development (early and delayed) of hemolysis after treatment are defined as follows:
  Early Hemolytic anemia is defined as 10% or greater decrease in hemoglobin levels and an increase of LDH levels to >390 U/L, or an increase of >= 10% above baseline occurring up to Day 8 of the study.
  Delayed hemolytic anemia might occur > 7 days after initiation of parenteral study drug (IV artesunate or IV cipargamin) during the study period. The event is characterized by a 10% or greater decrease in hemoglobin levels accompanied by increase of LDH levels to >390 U/L, or an increase of >= 10% compared to the values measured at Day 8 of the study.
Percentage of participants with neurological sequelae at Day 29 | Day 29
  Detailed neurological examination will be conducted and relevant medical history collected under the following categories to assess the extent of neurological signs and symptoms at baseline and to monitor the extent of neurological sequelae in follow-up visits:
  1. Consciousness
  2. Cranial Nerve Palsy
  3. Motor system
  4. Convulsions
  5. Sense organs (Examination more useful at time of hospital discharge and in follow-up visits)
Percentage of participants achieving at least 90% reduction in Plasmodium falciparum (P. falciparum) | Day 2 (24 hours), Day 3 (48 hours)
  A blood draw will be performed at each collection time point for parasitemia assessment
Time to parasite clearance (PCT) | Day 1 (12 hours), Day 2 (24 hours), Day 3 (48 hours) and Day 4 (72 hours)
  Parasite Clearance Time (PCT) is defined as the time from the first dose until the first total and continued disappearance of asexual parasite forms which remained at least a further 24 hours
Time to fever clearance (FCT) | Day 1 (12 hours), Day 2 (24 hours), Day 3 (48 hours) and Day 4 (72 hours)
  Fever Clearance Time (FCT) is defined as the time from the first dose until the first time the axillary body temperature decreased below and remained below 37.5°C axillary or 38.0°C oral/tympanic/rectal for at least a further 24 hours.
Percentage of participants achieving P. falciparum parasite reduction ratios (PRR) at 12, 24 and 48 hours | Day 1 (12 hours), Day 2 (24 hours) and Day 3 (48 hours)
  PRR is defined as the ratio of asexual parasite at baseline divided by asexual parasite at post-baseline. If the asexual parasite count at post-baseline is 0, the half value of detection limit will be used to calculate the ratio.
Percentage of participants with recrudescence and reinfection | Day 29
  Time to event (recrudescence or reinfection) will be calculated from the time of first study medication to the date of first event if a patient experiences the event and be censored at the time of last parasite assessment if a patient does not experience the event due to whatever reason.
  Reinfection is defined as appearance of asexual parasites after clearance of initial infection with a genotype different from those parasites present at baseline.
  Recrudescence is defined as appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at baseline.
  Reinfection and Recrudescence must be confirmed by PCR analysis.
Time to recover from prostration | Day 1 to Day 29
  To assess recovery of participants as measured by time (days and hours) to discharge from hospital or recovery from prostration compared to baseline.
Time to switch to oral therapy | Day 3 to Day 29
  Time to switch participants from IV therapy to Coartem (standard of drug for oral therapy) will be analyzed.
Time to discharge from hospital | Day 3 to Day 29
  All participants will be hospitalized. Time (Days and Hours) to discharge from hospital will be analyzed.
Number of Participants impacted on safety and tolerability assessments | Day 1 to Day 29
  Adverse events (AE), Serious Adverse events (SAEs) will be collected from first dosing, Death including whether in-hospital death and routine laboratory assessments will be done up to last follow-up visit or until the event has resolved to baseline grade or better or the event was assessed stable by the investigator or the participant was lost to follow-up or withdrew consent.
Observed maximum plasma concentration (Cmax) of IV Cipargamin | Day 1 - Day 8
  Blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) of IV Cipargamin | Day 1 - Day 8
  Blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of IV Cipargamin | Day 1 - Day 8
  Blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Area under the concentration time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) of IV Cipargamin | Day 1 - Day 8
  Blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-inf) will be listed and summarized using descriptive statistics.
Area Under the plasma concentration-time Curve from the time 0 to the last observed quantifiable concentration (AUC(0-t)) of IV Cipargamin | Day 1 - Day 8
  Blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-t) will be listed and summarized using descriptive statistics.
AUC(0-t) divided by the dose administered (AUC(0- t)/D) of IV Cipargamin | Day 1 - Day 8
  Blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-t)/D will be listed and summarized using descriptive statistics.
Terminal elimination half life (T^1/2) of IV Cipargamin | Day 1 - Day 8
  Blood samples will be collected for activity-based pharmacokinetics characterization. The half-live will be listed and summarized using descriptive statistics.
Total systemic clearance for intravenous administration (CL) of IV Cipargamin | Day 1 - Day 8
  Blood samples will be collected for activity-based pharmacokinetics characterization. CL will be listed and summarized using descriptive statistics.
volume of distribution during the terminal phase following intravenous elimination (Vz) of IV Cipargamin | Day 1 - Day 8
  Blood samples will be collected for activity-based pharmacokinetics characterization. Vz will be listed and summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Burkina Faso (2):
  - Novartis Investigative Site, Burkina Faso
  - Novartis Investigative Site, Ouagadougou
- Côte d’Ivoire (2):
  - Novartis Investigative Site, Abidjan
  - Novartis Investigative Site, Agboville
- Novartis Investigative Site, Kinsasha, Democratic Republic of Congo, Democratic Republic of the Congo
- Novartis Investigative Site, Siaya, Kenya
- Novartis Investigative Site, Manhiça, Maputo Province, Mozambique
- Novartis Investigative Site, Kigali, Rwanda
- Novartis Investigative Site, Tororo, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of participants who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com